CLINICAL TRIAL: NCT06172465
Title: Comparison of Bilateral Oblique Transversus Abdominis Plane Block (OSTAPB) and Bilateral External Oblique Intercostal Plane Block (EOIPB) in Laparoscopic Cholecystectomies
Brief Title: Comparison of OSTAP and EOIP Blocks in Laparoscopic Cholecystectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: trunk block
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Analgesia; Pain, Post Operative
Keywords: laparoscopic cholecystectomy; oblique subcostal transversus abdominis plane block; external oblique interfascial plane block
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: two interventional group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The anesthetist who will perform the blocks will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another anesthetist blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group external oblique intercostal plane block (Active Comparator): While patients are still under general anesthesia, external oblique intercostal block (EOIB) will be performed bilaterally according to appropriate asepsis/antisepsis rules at end of the surgery.
  Interventions: Other: EOIP
- group oblique subcostal transversus abdominis plane block (Active Comparator): Ultrasound-guided bilateral OSTAP block performed at end of the surgery. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed
  Interventions: Other: OSTAP

INTERVENTIONS:
Other: EOIP — Ultrasound guided External oblique intercostal block will be performed bilaterally.
  Arms: group external oblique intercostal plane block
Other: OSTAP — Ultrasound guided oblique subcostal transversus abdominis plane block will be performed bilaterally.
  Arms: group oblique subcostal transversus abdominis plane block

SUMMARY:
Laparoscopic cholecystectomy (LC) surgery causes postoperative severe pain. As part of multimodal analgesia aimed at reducing postoperative opioid consumption and providing effective analgesia, ultrasound (US)-guided transversus abdominis plane block (TAP) and external oblique intercostal plane block (EOIPB) will be applied as regional anesthesia methods. There is no study in the literature comparing OSTAP and EOIP blocks, and our goal is to evaluate the analgesic effectiveness between OSTAP and EOIP blocks in LC surgeries.

DETAILED DESCRIPTION:
Patients will be divided into two groups, and general anesthesia will be administered to all. Before extubation, one group will receive an external oblique intercostal nerve block, while the other group will receive an oblique subcostal transversus abdominis plane block. The randomization of the study will be carried out by a computer-generated randomization code (computer-generated) by a physician who will not be involved in patient follow-up. The interfascial plane block (either external oblique intercostal block or oblique subcostal block) will be provided to an anesthesiologist in a sealed envelope by an independent assistant staff member outside the study. The patient will not be aware of which block is applied. The anesthesiologist performing the block will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be conducted by another anesthesiologist unaware of the study.

For standardization, the block procedure will be performed by an experienced anesthesiologist who has completed at least 20 previous successful and uncomplicated procedures.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35 kg/m² Patients with ASA scores I and II

Exclusion Criteria:

* Patients who do not want to be included in the study Psychiatric and neurological disease with blurred consciousness Patients with ASA > 3 BMI > 35 kg/m² Abnormality in coagulation parameters History of allergy to local anesthetic drugs Infection at the injection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | up to 24 hours
  tramadol consumption in the first 24 hours after surgery

SECONDARY OUTCOMES:
NRS scores | At 1,3, 6, 12, 18, 24 hours
  NRS scores in the first 24 hours after surgery
Quality of recovery | 24 hours
  QR15 scores
Nausea and vomiting | At 1,3, 6, 12, 18, 24 hours
  Nausea and vomiting scores in the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: gamze MD ertaş, specialist, Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No